CLINICAL TRIAL: NCT04583709
Title: ECG Belt to Assess Electrical Synchronization in Patients With Left Bundle Branch Pacing and His-Purkinje Conduction System Optimized Cardiac Resynchronization Therapy (ECG Belt)
Brief Title: ECG Belt to Assess Electrical Synchronization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pugazhendhi Vijayaraman (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Pugazhendhi Vijayaraman, Sponsor-Investigator, Geisinger Clinic
Organization: Geisinger Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-0465
Record Dates: First submitted 2020-09-29; First posted 2020-10-12 (Actual); Results first posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-07

CONDITIONS: Bradycardia; Heart Failure
MeSH Terms: conditions — Bradycardia; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ECG Belt (Experimental): ECG belt will be used to record ECG during baseline rhythm, LBBP in unipolar and bipolar configurations and / or during HOT-CRT using HBP or LBBP. These ECG belt characteristics would then be compared with baseline and existing data on RV pacing and traditional Biventricular pacing.
  Interventions: Device: ECG Belt

INTERVENTIONS:
Device: ECG Belt — ECG Belt Research System Procedure LBBP Native conduction RV pacing if available Bipolar LBBP Unipolar LBBP - nonselective and selective (different outputs) Fusion pacing with native conduction at different Atrioventricular (AV) delays
  HOT-CRT Native conduction HBP / LBBP HOT-CRT AV delay optimization. Medtronic Device (pacemaker/ICD) based Holter recording during the ECG belt recording

SUMMARY:
The objective of the study is to assess the utility of ECG Belt to understand the conduction and ECG characteristics of Left Bundle Branch Pacing (LBBAP) and His-Optimized Cardiac Resynchronization Therapy (HOT-CRT) and compare with preexisting data in traditional Cardiac Resynchronization Therapy (CRT) and Right Ventricular Pacing (RVP).

DETAILED DESCRIPTION:
The objective of the study is to assess the utility of ECG Belt to understand the conduction and ECG characteristics of LBBP and HOT-CRT and compare with preexisting data in traditional CRT and RVP.

Specific Objective:

* To demonstrate and establish electrical resynchronization using ECG Belt Research System in Left Bundle Branch Pacing (LBBP) and HOT-CRT.
* To assess ECG Belt derived native conduction parameters and compare them to LBBP and HOT-CRT.
* To compare with historic ECG belt parameters obtained for right ventricular pacing/ Biventricular pacing in prior studies.

The ECG Belt study is a prospective, single-center, investigational, pre-market research study. The study team will identify all patients who satisfy the inclusion and exclusion criteria. The study team will evaluate the ECG Belt Research System to assess the electrical characteristics of conduction system pacing in patients with preexisting LBBP or HOT-CRT.

Eligible patients would have successfully undergone LBBP using Medtronic 3830 lead. LBBP will be confirmed at implant using left bundle potentials recorded from the lead, ECG morphology during unipolar and bipolar pacing, peak LV activation time and lead depth in the LV septum by contrast at implant and 2D echo post-implant.

ECG belt would be used to record ECG during baseline rhythm, LBBP in unipolar and bipolar configurations and / or during HOT-CRT using His-Bundle Pacing (HBP) or LBBP. These ECG belt characteristics would then be compared with baseline and existing data on Right Ventricular RV pacing and traditional Biventricular pacing.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years of age
2. Patient has a previously implanted LBBP lead for bradycardia indication or heart failure indication with one of the following at Geisinger within the last 5 years:

   * LBBP
   * LBBP+LV lead
   * HBP+LV
3. Patient is willing to comply with all study procedures and be available for the duration of the study.

Exclusion Criteria:

1. Inability to provide informed consent
2. Pregnant
3. Enrolled in a concurrent study that may confound the results of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pugazhendi Vijayaraman, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania, United States

REFERENCES:
- [Derived] Vijayaraman P, Hughes G, Manganiello M, Johns A, Ghosh S. Non-invasive assessment of ventricular electrical heterogeneity to optimize left bundle branch area pacing. J Interv Card Electrophysiol. 2023 Aug;66(5):1103-1112. doi: 10.1007/s10840-022-01315-9. Epub 2022 Jul 30. PMID 35907107

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients will be identified by clinician referrals, or by review of the electronic health record (EHR) of patients. Research staff will contact potential subjects and invite them to participate, either in clinic or by phone.
  First subject enrolled: 13 Jan 2021 Last subject enrolled: 18 Jun 2021 (follow up completed 25 Jun 2021)
Groups:
- ECG Belt: The ECG Belt Research System will be used to evaluate and assess the electrical characteristics of conduction system pacing in patients with preexisting LBBAP or HOT-CRT.
  ECG belt will be used to record ECG during baseline rhythm, LBBP in unipolar and bipolar configurations and / or during HOT-CRT using HBP or LBBP. These ECG belt characteristics would then be compared with baseline and existing data on RV pacing and traditional Biventricular pacing.
  ECG Belt: ECG Belt Research System Procedure All patients will share the same recruitment process, inclusion and exclusion criteria and same procedures. Patients are allocated to ECG Belt group and data will be collected according to their preexisting therapy.
  Data includes:
  LBBP Native conduction RV pacing if available Bipolar LBBP Unipolar LBBP - nonselective and selective (different outputs) Fusion pacing with native conduction at different Atrioventricular (AV) delays
  HOT-CRT Native conduction HBP / LBBP HOT-CRT AV delay optimization. Medtronic Device (pacemaker/ICD) based Holter recording during the ECG belt recording
Period: Overall Study
Arm/Group | ECG Belt
Started (Initial enrollment) | 20
Completed (Completion of study participation of last enrollment (patient 20)) | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- ECG Belt: ECG belt will be used to record ECG during baseline rhythm, LBBP in unipolar and bipolar configurations and / or during HOT-CRT using HBP or LBBP. These ECG belt characteristics would then be compared with baseline and existing data on RV pacing and traditional Biventricular pacing.
  ECG Belt: ECG Belt Research System Procedure LBBP Native conduction RV pacing if available Bipolar LBBP Unipolar LBBP - nonselective and selective (different outputs) Fusion pacing with native conduction at different Atrioventricular (AV) delays
  HOT-CRT Native conduction HBP / LBBP HOT-CRT AV delay optimization. Medtronic Device (pacemaker/ICD) based Holter recording during the ECG belt recording
Arm/Group | ECG Belt
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: • ECG Belt Analysis of Standard Deviation of Activation Times (SDAT) of LBBP Compared to Native Conduction
Description: Change in SDAT following LBBP measured in ms using ECG Belt
Time Frame: Visit 1 Baseline-50 minutes
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | ECG Belt
Number analyzed (Participants) | 20
ms
  SDAT at Baseline | 38.6 (9.03)
  SDAT at Optimized LBBAP | 20.5 (7.54)

2. Primary Outcome: • ECG Belt Analysis of Left Ventricular Activations Times (LVAT) of LBBP Compared to Baseline
Description: Change in LV activation times measured in ms using ECG Belt
Time Frame: Visit 1 Baseline-50 minutes
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | ECG Belt
Number analyzed (Participants) | 20
ms
  LVAT at Baseline | 61.4 (21)
  LVAT at Optimized LBBAP | 44.4 (4.3)

3. Primary Outcome: • ECG Belt Analysis of QRS Duration at Baseline Compared to Various LBBP Options
Description: Change in QRS duration measured in ms using ECG Belt
Time Frame: Visit 1 Baseline-50 minutes
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | ECG Belt
Number analyzed (Participants) | 20
ms
  QRSd at Baseline | 152 (24)
  QRSd at Optimized LBBAP | 133 (20)

4. Primary Outcome: • ECG Belt Analysis of LV Dispersion of HOT-CRT Compared to Baseline
Description: LV dispersion measured using ECG Belt
Time Frame: Visit 1 Baseline- 50 minutes
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | ECG Belt
Number analyzed (Participants) | 20
ms
  LV dispersion at Optimized LBBAP | 11.6 (11.64)
  LV dispersion at Baseline | 29.5 (15.01)

5. Primary Outcome: • ECG Belt Analysis of RV Dispersion of HOT-CRT Compared to Baseline
Description: RV dispersion measured using ECG Belt
Time Frame: Visit 1 Baseline- 50 minutes
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | ECG Belt
Number analyzed (Participants) | 20
ms
  RV dispersion at Optimized LBBAP | 21.1 (7.84)
  RV dispersion at Baseline | 42.5 (9.31)

ADVERSE EVENTS:
Time Frame: Study related adverse events were collected during the one year time span of enrollment and follow up. For each participant, adverse event data was collected during their time participating in the study (1 week).
Description: Patients will be asked about adverse events related to the use of the ECG Belt. These data will not be monitored in real time and patients will be educated on the need to contact their physician directly should they have any medical concern.
  Only ECG Belt related SAE/AE's will be collected and reported and then assessed if it is device related.
Arm/Group | ECG Belt
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ECG Belt (N=20)
Product related adverse event (Product Issues) | 1 (1) — Redness on skin under electrodes of ECG Belt system

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/09/NCT04583709/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT04583709/ICF_001.pdf